CLINICAL TRIAL: NCT01066546
Title: An Open-Label Extension To The B1451006 Protocol To Evaluate The Safety And Efficacy Of Dimebon (Latrepirdine, PF-01913539) In Subjects With Moderate-To-Severe Alzheimer's Disease
Brief Title: An Extension To The B1451006 Protocol To Evaluate The Safety and Efficacy of Dimebon In Subjects With Moderate-to-Severe Alzheimer's Disease
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: See termination reason in detailed description.
Sponsor: Pfizer (Industry)
Collaborators: Medivation, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B1451030
Record Dates: First submitted 2010-02-09; First posted 2010-02-10 (Estimated); Results first posted 2012-10-02 (Estimated); Last update posted 2012-10-02 (Estimated); Status verified 2012-08

CONDITIONS: Alzheimer's Disease
Keywords: Delirium; Dementia; Amnestic; Cognitive Disorders; Mental Disorders; Nervous System Diseases; Central Nervous System Diseases
MeSH Terms: conditions — Alzheimer Disease; Delirium; Dementia; Cognitive Dysfunction; Mental Disorders; Nervous System Diseases; Central Nervous System Diseases | interventions — latrepirdine; Administration, Oral

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Dimebon (Experimental)
  Interventions: Drug: Dimebon tablet for oral administration

INTERVENTIONS:
Drug: Dimebon tablet for oral administration — 10 mg TID for Week 1, followed by 20 mg TID for remainder of study

SUMMARY:
The purpose of this study is to evaluate the long-term safety and tolerability of dimebon in subjects with moderate-to-severe Alzheimer's Disease.

DETAILED DESCRIPTION:
This study was terminated on May 7, 2010 due to modification of the dimebon development plan, following the lack of demonstration of efficacy in the completed DIM14 (CONNECTION) Study. The study was not terminated due to any safety findings. Dimebon has been well-tolerated in clinical trials. Demonstration of efficacy for dimebon in Alzheimer's disease is pending completion of the ongoing DIM18 (CONCERT) Study.

ELIGIBILITY:
Inclusion Criteria:

* Successful completion of 6 months treatment in the previous B1451006 Phase 3 dimebon study

Exclusion Criteria:

* Any major medical illness or unstable medical condition that may increase the risk associated with study participation or investigational product administration or may interfere with the ability to interpret study safety data

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2010-04; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (5):
- United States (5):
  - Pfizer Investigational Site, Costa Mesa, California
  - Pfizer Investigational Site, Encino, California
  - Pfizer Investigational Site, Los Alamitos, California
  - Pfizer Investigational Site, Newport Beach, California
  - Pfizer Investigational Site, Delray Beach, Florida

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1451030&StudyName=An%20Extension%20To%20The%20B1451006%20Protocol%20To%20Evaluate%20The%20Safety%20and%20Efficacy%20of%20Dimebon%20In%20Subjects%20With%20Moderate-to-Severe%20Alzheimer%27s%20D

RESULTS

PARTICIPANT FLOW:
Groups:
- Dimebon: Dimebon (latrepirdine) 10 milligram (mg) tablet orally three times a day for 1 week (titration period), followed by dimebon (latrepirdine) 20 mg tablet orally three times a day. Treatment was administered until participant withdrawal or study termination.
Period: Overall Study
Arm/Group | Dimebon
Started | 5
Completed | 0
Not Completed | 5
Not completed — Study terminated by sponsor | 5

BASELINE CHARACTERISTICS:
Groups:
- Dimebon: Dimebon (latrepirdine) 10 mg tablet orally three times a day for 1 week (titration period), followed by dimebon (latrepirdine) 20 mg tablet orally three times a day. Treatment was administered until participant withdrawal or study termination.
Arm/Group | Dimebon
Number analyzed (Participants) | 5
Age, Customized [Number; unit: participants]
  Less than 50 years | 0
  50 to 59 years | 1
  60 to 69 years | 0
  70 to 79 years | 1
  80 to 85 years | 2
  Greater than 85 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs)
Description: An adverse event is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship.
Time Frame: Baseline up to 4 weeks after last dose of study treatment
Population: Safety analysis population included all enrolled participants who received at least 1 dose of study treatment, including partial doses.
Measure: Number; unit: participants
Arm/Group | Dimebon
Number analyzed (Participants) | 5
participants | 2

2. Secondary Outcome: Change From Baseline in Severe Impairment Battery (SIB) at Week 6, 12 and 26
Description: SIB developed for evaluation of cognitive function in participants, who demented to a degree that they cannot complete conventional neuropsychological testing. Test items consisted of simple, one-step commands presented with gestural cues and instructions that were repeated if necessary. SIB test consisted of 51-item scale, divided into 9 subscales: social interaction (0-6), memory (0-14), orientation (0-6), language (0-46), attention (0-6), praxis (0-8), visuospatial ability (0-8), construction(0-4), orienting to name(0-2). Total possible score:0-100; lower score=greater cognitive impairment.
Time Frame: Baseline, Week 6, 12, 26
Population: Data was not analyzed due to early termination of study and no participants completed the pre-defined visit schedule.
Arm/Group | Dimebon
Number analyzed (Participants) | 0

3. Secondary Outcome: Change From Baseline in Alzheimer's Disease Cooperative Study-Activities of Daily Living-Severe Version (ADCS-ADLsev) at Week 6, 12 and 26
Description: ADCS-ADLsev: 19-item scale measures basic and instrumental abilities in participant population and had good metric properties and reliability in detecting change. Individual score range: 0 to 5 for telephone, 0 to 4 for dressing, watch television, get around outside home, 0 to 3 for eating, walking, toilet, bathing, grooming, conversation/small talk, clear dishes, find personal belongings, obtain beverages, dispose of garbage, left on own, 0 to 1 for run water from and turn off faucet to wash hands, turn on and off light. Total score range: 0 to 54 lower scores=greater functional impairment.
Time Frame: Baseline, Week 6, 12, 26
Population: Data was not analyzed due to early termination of study and no participants completed the pre-defined visit schedule.
Arm/Group | Dimebon
Number analyzed (Participants) | 0

4. Secondary Outcome: Change From Baseline in Mini-Mental State Examination (MMSE) at Week 12 and 26
Description: MMSE measured general cognitive functioning: orientation, memory, attention, concentration, naming, repetition, comprehension, and ability to create a sentence and to copy two intersecting polygons. Total score derived from sub-scores; ranged from 0 to 30, higher score indicates better cognitive state.
Time Frame: Baseline, Week 12, 26
Population: Data was not analyzed due to early termination of study and no participants completed the pre-defined visit schedule.
Arm/Group | Dimebon
Number analyzed (Participants) | 0

5. Secondary Outcome: Change From Baseline in Neuropsychiatric Inventory (NPI) at Week 6, 12 and 26
Description: NPI:12-domain caregiver assessment of behavioral disturbances occurring in dementia: delusions, hallucinations, agitation/aggression, depression/dysphoria, anxiety, elation/euphoria, apathy/indifference, disinhibition, irritability/lability, motor disturbance, appetite/eating, nighttime behavior. Severity(1=Mild to 3=Severe),frequency(1=occasionally to 4=very frequently) scales recorded for each domain; frequency*severity=each domain score(range 0-12). Total score=sum of each domain score(range 0-144);higher score=greater behavioral disturbances;negative change score from baseline=improvement.
Time Frame: Baseline, Week 6, 12, 26
Population: Data was not analyzed due to early termination of study and no participants completed the pre-defined visit schedule.
Arm/Group | Dimebon
Number analyzed (Participants) | 0

6. Secondary Outcome: Sum of Delusions and Hallucinations Sub-domain Scores of Neuropsychiatric Inventory (NPI) at Week 26
Description: NPI is a 12-domain caregiver assessment of behavioral disturbances occurring in dementia. Severity (1=Mild to 3=Severe) and frequency (1=occasionally to 4=very frequently) scales were recorded separately for each domain and their product gives individual domain score (range 0-12). Sum of delusions and hallucinations sub-domain scores of NPI was calculated as a measure of Alzheimer's Disease (AD) related psychosis. Total possible score range: 0-24 with higher score indicating greater behavioral disturbances.
Time Frame: Week 26
Population: Data was not analyzed due to early termination of study and no participants completed the pre-defined visit schedule.
Arm/Group | Dimebon
Number analyzed (Participants) | 0

7. Secondary Outcome: Change From Baseline in Resource Utilization in Dementia - Lite Version (RUD-Lite) at Week 12 and 26
Description: RUD Lite: instrument used to assess amount of both formal and informal resources used by demented participants and primary caregiver. It was completed by caregivers and compiles data on following resources: use of social services, frequency and duration of hospitalizations, all contacts with health care professionals, participant living accommodations, amount of time the caregiver spends giving care and the impact of care giving on the caregiver's job. Overall cost of care was evaluated to quantify the resources utilized.
Time Frame: Baseline, Week 12, 26
Population: Data was not analyzed due to early termination of study and no participants completed the pre-defined visit schedule.
Arm/Group | Dimebon
Number analyzed (Participants) | 0

8. Secondary Outcome: Change From Baseline in European Quality of Life 5 Domain Scale (EQ-5D) at Week 12 and 16
Description: EQ-5D: participant rated questionnaire to assess health-related quality of life in terms of a single utility score. Health State Profile component assesses level of current health for 5 domains: mobility, self-care, usual activities, pain and discomfort, and anxiety and depression; 1 indicates better health state (no problems); 3 indicates worst health state ("confined to bed"). Total possible score is sum of individual items, ranged from 5 to 15; lower score indicated a better health state.
Time Frame: Baseline, Week 12, 26
Population: Data was not analyzed due to early termination of study and no participants completed the pre-defined visit schedule.
Arm/Group | Dimebon
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Dimebon
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 2/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dimebon (N=5)
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Urinary tract infection (Infections and infestations) | 1

LIMITATIONS AND CAVEATS:
Results are not summarized because of early termination of the study due to modification in the development plan of the study treatment following lack of demonstration of efficacy in the completed DIM14 CONNECTION (B1451002/NCT00675623) study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.